CLINICAL TRIAL: NCT05490407
Title: ATP7A Transporter as Biomarker for Predicting Chemoresistance of Serous Ovarian Cancer
Brief Title: Role of the ATP7A Transporter in Ovarian Cancer
Acronym: ATHOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine, Institute of Pharmacology and Experimental Toxicology (Unknown)
Responsible Party: Principal Investigator, David Lukanovic, Asist. David Lukanovic, MD, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UMCL
Record Dates: First submitted 2021-05-11; First posted 2022-08-05 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Gynecologic Cancer; Ovarian Cancer; High Grade Serous Carcinoma; Chemotherapy Effect
Keywords: Ovarian cancer; Chemoresistance; Predictive marker; ATP7A
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HGSOC (Other): high-grade serous ovarian cancer patients (FIGO stages III and IV) with ascites, for whom neoadjuvant chemotherapy is recommended.
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — Patients will receive neoadjuvant chemotherapy according to ESGO guidelines

SUMMARY:
Ovarian cancer has the highest mortality rate among all gynecologic cancers, with most patients presenting with advanced stage tumors. About a third of patients do not respond to primary platinum-based chemotherapy treatment, and over time up to 80 % of others develop chemoresistance, rendering recurrent disease incurable. Despite all the studies published in the literature, it has not been proven that the number of cells with expressed ATP7A in certain tumors increases independently of the therapy. In addition, no study has been conducted on a sample of patients with confirmed serous histology of ovarian cancer only. The aim of the study is to demonstrate increased expression of the ATP7A transporter in cells resistant to carboplatin.

DETAILED DESCRIPTION:
RATIONALE:

Recent studies suggest that the copper efflux transporters ATP7A plays an important role in platinum resistance. Despite all the studies published in the literature, it has not been proven that the number of cells with expressed ATP7A in certain tumors increases independently of the therapy. In addition, no study has been conducted on a sample of patients with confirmed serous histology of ovarian cancer only. The literature concludes that new methods are required to detect resistant tumor cells at an early chemotherapy stage and suitably adapt treatment. There is still much uncertainty regarding how the fate of platinum compounds in a cell follows the regulatory copper pathways, especially during transport from the cell. The question is also to what extent these processes are cell-specific, especially because experiments to date regarding the role of ATP7A in resistance to platinum compounds have been conducted on nonserous cell lines (especially of the endometrioid histological type).

AIM OF THE STUDY:

Study will evaluate the ATP7A transporter as an important mediator of chemoresistance to platinum compounds to obtain an additional criterion for the optimal treatment strategy for serous ovarian cancer patients. The focus will primarily be on intrinsic chemoresistance, which determines the initial response to chemotherapy. Research to date has failed to evaluate the influence of ATP7A transporter expression solely on serous ovarian cancer.

The study will demonstrate increased expression of the ATP7A transporter in cells resistant to carboplatin. Because the measurement of ATP7A in bodily fluids is unreliable, the plan is to measure ceruloplasmin in the patients' ascites. Ceruloplasmin is the main copper-transporting protein in the blood. It is synthesized in the cell and, according to findings in the literature, it is ATP7A that is responsible for delivering copper to ceruloplasmin. When copper binds to ceruloplasmin, there is no other way for it to cross the plasma membrane than via the ATP7A transporter. By measuring the ceruloplasmin level in the ascites, ATP7A activity or its localization on the plasma membrane could indirectly be measured as well. To confirm the suitable measurement of ceruloplasmin in the ascites, its values in the patients' blood plasma and tissue will be measured.

METHODS:prospective clinical trial It will include 30 high-grade serous ovarian cancer patients (FIGO stages III and IV) with ascites. The patients will be presented to the gynecological-oncological consultation team at the Ljubljana Division of Gynecology and Obstetrics. Patients for whom neoadjuvant chemotherapy is recommended will be included in the trial.

STATISTICAL ANALYSES: The normality of numerical variables' distribution will be tested with the Shapiro-Wilk test. Relevant parametric tests (Student's t-test) or nonparametric tests (the two-tailed Mann-Whitney U-test) will be used to compare groups.

ELIGIBILITY:
Inclusion Criteria:

* high-grade serous ovarian cancer patients (FIGO stages III and IV) with ascites, for whom neoadjuvant chemotherapy is recommended

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
concentration of ceruloplasmin | before the start of neoadjuvant chemotherapy
  To measure concentration of ceruloplasmin in blood and ascites
expression of ATP7A | before the start of neoadjuvant chemotherapy
  To measure expresion of ATP7A

SECONDARY OUTCOMES:
concentration of ceruloplasmin after chemotherapy | after neoadjuvant chemotherapy - within 6 months
  To measure concentration of ceruloplasmin after three to six chemotherapy cycles
expresion of ATP7A after chemotherapy | after neoadjuvant chemotherapy - within 6 months
  To measure expresion of ATP7A after three-six cycles of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Borut Kobal, MD; PhD, Study Director — Department of Gynecology, Division of Gynecology and Obstetrics, Ljubljana University Medical Center; Katarina Černe, MD, PhD, Study Chair — Institute of Pharmacology and Experimental Toxicology, Medical Faculty, University Ljubljana
Locations (2):
- Slovenia (2):
  - Department of Gynecology, Division of Gynecology and Obstetrics, Ljubljana University Medical Center, Ljubljana
  - Institute of Pharmacology and Experimental Toxicology, Faculty of Medicine, University of Ljubljana., Ljubljana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lukanovic D, Herzog M, Kobal B, Cerne K. The contribution of copper efflux transporters ATP7A and ATP7B to chemoresistance and personalized medicine in ovarian cancer. Biomed Pharmacother. 2020 Sep;129:110401. doi: 10.1016/j.biopha.2020.110401. Epub 2020 Jun 20. PMID 32570116
- [Background] Colombo N, Sessa C, du Bois A, Ledermann J, McCluggage WG, McNeish I, Morice P, Pignata S, Ray-Coquard I, Vergote I, Baert T, Belaroussi I, Dashora A, Olbrecht S, Planchamp F, Querleu D; ESMO-ESGO Ovarian Cancer Consensus Conference Working Group. ESMO-ESGO consensus conference recommendations on ovarian cancer: pathology and molecular biology, early and advanced stages, borderline tumours and recurrent diseasedagger. Ann Oncol. 2019 May 1;30(5):672-705. doi: 10.1093/annonc/mdz062. PMID 31046081
- [Background] Samimi G, Safaei R, Katano K, Holzer AK, Rochdi M, Tomioka M, Goodman M, Howell SB. Increased expression of the copper efflux transporter ATP7A mediates resistance to cisplatin, carboplatin, and oxaliplatin in ovarian cancer cells. Clin Cancer Res. 2004 Jul 15;10(14):4661-9. doi: 10.1158/1078-0432.CCR-04-0137. PMID 15269138
- [Background] Samimi G, Varki NM, Wilczynski S, Safaei R, Alberts DS, Howell SB. Increase in expression of the copper transporter ATP7A during platinum drug-based treatment is associated with poor survival in ovarian cancer patients. Clin Cancer Res. 2003 Dec 1;9(16 Pt 1):5853-9. PMID 14676106
- [Background] Lukanović D, Kobal B, Černe K. Ovarian Cancer: Treatment and Resistance to Pharmacotherapy. Reproductive Medicine. 2022; 3(2):127-140. https://doi.org/10.3390/reprodmed3020011